CLINICAL TRIAL: NCT01583309
Title: Effects of Convective Therapies in Dialysis Patients
Acronym: ECTDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A. Manzoni Hospital (Other)
Responsible Party: Principal Investigator, Prof. Francesco Locatelli, Professor Francesco Locatelli, A. Manzoni Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONVESTUDY
Record Dates: First submitted 2012-04-17; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Uremia
Keywords: blood pressure; cardiovascular instability; symptomatic hypotension; online hemofiltration; online hemodiafiltration
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- low-flux hemodialysis (No Intervention)
- online pre-dilution hemofiltration (Experimental)
  Interventions: Procedure: online pre-dilution hemofiltration
- online pre-dilution hemodiafiltration (Experimental)
  Interventions: Procedure: online pre-dilution hemodiafiltration

INTERVENTIONS:
Procedure: online pre-dilution hemofiltration — Online pre-dilution hemofiltration was performed with a synthetic high-flux membrane and an infusate/blood flow ratio of one
  Other Names: online pre-dilution hemofiltration Technique
  Arms: online pre-dilution hemofiltration
Procedure: online pre-dilution hemodiafiltration — Online pre-dilution hemodiafiltration was performed with a synthetic high-flux membrane with an infusate/blood flow ratio of 0.6 and a dialysate plus infusate rate of 700 ml/min.
  Other Names: online pre-dilution hemodiafiltration Technique
  Arms: online pre-dilution hemodiafiltration

SUMMARY:
Convective therapies have been proposed for improving chronic dialysis patient outcomes, including intradialytic symptomatic hypotension.

To evaluate the frequency of sessions with intradialytic symptomatic hypotension in different types and doses of convective therapies compared with low-flux hemodialysis (HD), the investigators performed a multicentre, open-label, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients aged 18-80 years
* thrice-weekly HD or HDF for at least 6 months
* body weight less or equal to 90 Kg
* stable clinical condition
* written consent

Exclusion Criteria:

* infections
* malignancies
* active systemic diseases
* active hepatitis or cirrhosis
* unstable diabetes
* diuresis higher than 200 ml/24h
* dysfunction of vascular access
* blood flow rate less than 300 ml/min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2003-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Intradialytic symptomatic hypotension | all dialysis sessions, three per week, for 2 years
  Intradialytic symptomatic hypotension was defined as a rapid symptomatic fall of the systolic blood pressure by at least 30 mmHg or that required nursing and/or medical intervention

SECONDARY OUTCOMES:
Resistance to erythropoiesis-stimulating agents | Monthly for 2 years
  Resistance to erythropoiesis-stimulating agents was measured as (EPO therapy in IU/week)/(Hb in g/dL*body wheight in kg)
Calcium-phosphate metabolism | Monthly for 2 years
  Outcome measures: phosphatemia, calcemia and PTH
Beta2 microglobulin | Every six months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Locatelli, Professor, Study Chair — A. Manzoni Hospital, Lecco - Italy
Locations (27):
- Italy (27):
  - Ospedale S.Marta S.Venera, Acireale (CT)
  - Ospedale F. Miulli, Acquaviva delle Fonti
  - Ospedale Civile, Alghero
  - Ospedale regionale di Aosta, Aosta
  - Ospedale degli Infermi, Biella
  - Ospedale SS. Trinità ASL 8, Cagliari
  - S. Michele Hospital, Cagliari
  - Ospedale Civile "P. Merlo", La Maddalena
  - Alessandro Manzoni Hospital, Lecco
  - Ospedale "C. POMA", Mantova
  - T. EVOLI, Melito di Porto Salvo
  - Ospedale dell'Angelo, Mestre
  - Policlinico Multimedica IRCCS, Milan
  - Federico II, Napoli
  - Ospedale San Francesco, Nuoro
  - San Giovanni di Dio, Olbia
  - Ospedale Antonio Segni, Ozieri
  - Ospedale Maggiore, Parma
  - Fondazione Maugeri, Pavia
  - Ospedale " E. AGNELLI ", Pinerolo
  - Dipartimento territoriale ASL 8, Quartu Sant'Elena
  - Ospedale S.Maria delle Croci, Ravenna
  - Azienda Ospedaliera "Bianchi Melacrino Morelli,", Reggio Calabria
  - Ospedale Bolognini, Seriate
  - Ospedale Agostino Landolfi, Solofra
  - Ospedale San Camillo, Sorgono
  - ASL 2 Olbia - P.O. "P. Dettori",, Tempio Pausania

REFERENCES:
- [Background] Bolasco P, Altieri P, Andrulli S, Basile C, Di Filippo S, Feriani M, Pedrini L, Santoro A, Zoccali C, Sau G, Locatelli F. Convection versus diffusion in dialysis: an Italian prospective multicentre study. Nephrol Dial Transplant. 2003 Aug;18 Suppl 7:vii50-4; discussion vii59-62. doi: 10.1093/ndt/gfg1080. PMID 12953031
- [Result] Locatelli F, Altieri P, Andrulli S, Bolasco P, Sau G, Pedrini LA, Basile C, David S, Feriani M, Montagna G, Di Iorio BR, Memoli B, Cravero R, Battaglia G, Zoccali C. Hemofiltration and hemodiafiltration reduce intradialytic hypotension in ESRD. J Am Soc Nephrol. 2010 Oct;21(10):1798-807. doi: 10.1681/ASN.2010030280. Epub 2010 Sep 2. PMID 20813866
- [Derived] Locatelli F, Altieri P, Andrulli S, Sau G, Bolasco P, Pedrini LA, Basile C, David S, Gazzanelli L, Tampieri G, Isola E, Marzolla O, Memoli B, Ganadu M, Reina E, Bertoli S, Ferrara R, Casu D, Logias F, Tarchini R, Mattana G, Passaghe M, Fundoni G, Villa G, Di Iorio BR, Pontoriero G, Zoccali C. Phosphate levels in patients treated with low-flux haemodialysis, pre-dilution haemofiltration and haemodiafiltration: post hoc analysis of a multicentre, randomized and controlled trial. Nephrol Dial Transplant. 2014 Jun;29(6):1239-46. doi: 10.1093/ndt/gfu031. Epub 2014 Feb 20. PMID 24557989